CLINICAL TRIAL: NCT03607773
Title: Mindfulness Group Intervention for Newly Diagnosed Persons With Multiple Sclerosis: A Pilot Study
Brief Title: Mindfulness for Newly Diagnosed Multiple Sclerosis
Acronym: MIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Morrow (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor-Investigator, Sarah Morrow, MS Specialist, Associate Professor, Primary Investigator, London Health Sciences Centre
Organization: London Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111561
Record Dates: First submitted 2018-07-12; First posted 2018-07-31 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Mindfulness
MeSH Terms: conditions — Multiple Sclerosis | interventions — Population Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI will not know which group each participant has been randomized to, nor will the study coordinator.
  One study team member, who is leading the Mindfulness sessions, will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Behavioural Intervention (MBI) group (Active Comparator): 10 one-hour mindfulness sessions
  Interventions: Behavioral: Mindfulness Behavioural Intervention (MBI) group
- Control group (No Intervention): Standard of care.

INTERVENTIONS:
Behavioral: Mindfulness Behavioural Intervention (MBI) group — While every MBI session is different, in general they will help you develop skills in focused attention, and emotional and behavioural regulation in a group environment made up of other people with MS who may share common experiences with you. MBI sessions are group-based which means you will be attending the sessions with other people who are also in this study and facilitated by trained personnel .
  Arms: Mindfulness Behavioural Intervention (MBI) group

SUMMARY:
Multiple Sclerosis (MS) is a chronic neurological disease often diagnosed in a person's 20s or 30s, at a time when most people are starting careers and families. In relapsing remitting (RR) MS new neurological symptoms suddenly develop over hours to days during relapses, and they do not start to resolve for days to weeks. Relapse symptoms may not completely disappear, such that disability accumulates over time. Further, most persons with RRMS will enter a progressive phase years after diagnosis. It is unpredictable when the transition to the progressive phase will occur and how quickly this progression will happen. Thus, receiving an MS diagnosis is a highly stressful event. Persons with MS (PwMS) often suffer from mood symptoms, which can further impair quality of life (QOL).

PwMS need support and the skills to effectively cope with the distress that comes with the uncertainty of a new MS diagnosis, as well as to minimize or prevent the onset of negative mood symptoms. One promising approach is mindfulness - a mental state of paying attention with intention, and accepting the present moment as it is without judgment. Scientific evidence supports the use of mindfulness based interventions (MBIs) in other chronic diseases to reduce stress, anxiety and depression, leading to improved physical function and QOL. MBIs decreased stress-related symptoms and the levels of stress hormones in the blood. As such, MBIs have the potential to lessen the negative consequences of stress in newly diagnosed PwMS.

DETAILED DESCRIPTION:
The investigators aim to assess if an MBI can reduce the negative impact of an MS diagnosis by improving coping skills. The investigator predicts that it will reduce perceived stress as well as stress markers in the blood, thus increasing overall QOL for newly diagnosed PwMS.

In this study, the investigator will randomly assign newly diagnosed PwMS to either MBI or standard treatment. The investigator administers the MBI under the format of the Mindfulness Ambassador Council (MAC), which was developed by the non-profit organization, Mindfulness Without Borders (MWB, www.mindfulnesswithoutborders.org). This intervention will consist of group meetings led by a mindfulness coach once a week for an hour over 10 weeks. We will include in the study PwMS that have been diagnosed with RRMS within the last year. We will assess measures of coping, mood symptoms and QOL before the intervention, after 10 weeks (or equivalent time for the standard treatment group) and then again 6 months later, to ensure any benefit continues over time.

First and foremost, PwMS will benefit from this type of research. This project could lead to a non-pharmacological, cost-effective intervention to help cope with the uncertainty that comes with an MS diagnosis as well as improves mood symptoms, psychosocial functioning and QOL, currently and over the long-term.

Sharing the results of this study will be a priority for us. We will present our results at national and international meetings as well as submit for journal publication. We will share our findings with other health care practitioners and with the lay public through community presentations and possible media releases.

ELIGIBILITY:
Inclusion Criteria:

1. Recently diagnosed with RRMS;
2. Must be within 1 year of an RRMS diagnosis at the time of the first MBI session;
3. Between 18-59 years of age inclusive; and
4. Fluent in English.

Exclusion Criteria:

1. Have bipolar disorder, schizophrenia, post-traumatic stress disorder, dissociation disorders or untreated depression or other psychiatric disease (at the PI's discretion) that could affect the study outcomesa major psychiatric disease such as bipolar disorder, schizophrenia or untreated severe major depressive disorder;
2. Use of marijuana more than 3x per week, or have other substance abuse, as determined by the PI;
3. Diagnosed with other neurological disorder(s) that would prevent participation in the intervention; or
4. Unable to attend at least 80% (8 of 10) of the MBI sessions (missing more than 20% of the sessions will result in removal from the study).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Change in coping skills | Within 1 month Pre-MBI sessions; Within 1 month Post-MBI sessions; 6 months post-MBI sessions.
  Brief COPE measure - was developed to assess a broad range of coping responses.28 questions with a 1-4 point scale for a total range of 28-116 with a lower score indicating better coping skills.
  This will be assessed at three time points and then aggregated to arrive at one reported value that represents "change in coping skills". This is indicated as an integer. Ex. Pre-MBI = 70 and Post-MBI = 50 and 6mo Post-MBI = 50 then the aggregated score would be -20.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Morrow, M.D., Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No